CLINICAL TRIAL: NCT03315273
Title: Measuring Motor Imagery Ability in Patients With Traumatic Brain Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2017/0826
Record Dates: First submitted 2017-10-03; First posted 2017-10-20 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Traumatic Brain Injury; Healthy
Keywords: Traumatic brain injury, motor imagery ability, validation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Comparison of 2 groups: one existing of patients with traumatic brain injury and one control group of healthy volunteers matched for age, sex and educational level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traumatic brain injury (Experimental): Patients who have suffered a traumatic brain injury will be assessed with a test battery including
  * a motor imagery ability questionnaire (MIQ-rs)
  * a mental rotation test
  * a chronometry test (TDMI)
  Interventions: Other: Test battery to measure the motor imagery ability
- Control (Active Comparator): Healthy volunteers matched for age, sex and educational level will be assessed with the same test battery including
  * a motor imagery ability questionnaire (MIQ-RS)
  * a mental rotation test
  * a chronometry test (TDMI)
  Interventions: Other: Test battery to measure the motor imagery ability

INTERVENTIONS:
Other: Test battery to measure the motor imagery ability — Participants will perform 3 different tests to measure the motor imagery ability

SUMMARY:
1. Validation of translated Motor Imagery ability questionnaire MIQ-RS
2. Investigating the Motor Imagery ability in patients with traumatic brain injury

DETAILED DESCRIPTION:
1. Translation of the MIQ-RS following the WHO guidelines. Followed by a validation of this translated questionnaire in patients with traumatic brain injury and in healthy volunteers.
2. Investigating the motor imagery ability using 3 different test

   * MIQ-RS (movement imagery questionnaire)
   * TDMI (time dependent motor imagery)
   * mental chronometry test

Patients and controls will perform all 3 test twice with an interval of 2 weeks to measure the test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* TBI minimum 3 months ago and maximal 1 year ago

Exclusion Criteria:

* Other neurological disorders
* Severe cognitive deficits, unable to understand the study protocol
* Severe motor impairment, unable to perform the TDMI (Time Dependent Motor Imagery) screening test

Control group:

Matched for age, sex and educational level No neurological disorders present

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Motor imagery ability | 2 assessments with an interval of 2 weeks
  Results of test battery assessing motor imagery ability
Validity translated MIQ-RS | 2 assessments with an interval of 2 weeks
  Validity of the translated MIQ-RS in patients with traumatic brain injury and healthy volunteers

SECONDARY OUTCOMES:
Test-retest reliability | 2 assessments with an interval of 2 weeks
  Test- retest reliability of the motor imagery ability test battery

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Oostra, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium